CLINICAL TRIAL: NCT05164783
Title: Multicenter Implementation of E-monitoring in Parkinson's Disease
Acronym: EPD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zuyderland Medisch Centrum (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Principal Investigator, Gerrit Tissingh, Dr. G. Tissingh, neurologist, Zuyderland Medisch Centrum
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Z2021125
Record Dates: First submitted 2021-10-28; First posted 2021-12-21 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Telemonitoring; Cost effectiveness; Quality of care; eHealth
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Implementation study with stepwise approach
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants (Experimental): Intervention: use of SCP
  Interventions: Combination Product: Sanacoach Parkinson (SCP)

INTERVENTIONS:
Combination Product: Sanacoach Parkinson (SCP) — A web-based monitoring tool for patients with PD, using questionnaires. It includes nine parts: 1) A 89-question, quarterly questionnaire about PD-symptoms. 2) Questionnaire responses are converted to scores on 16 PD-related domains. Both the current score and the score's change compared to the previous questionnaire are visible. 3) An interim evaluation is sent after 6 weeks with questions on any domains where a patient indicated problems. 4) A medication monitor can be initialized by the treating physician to evaluate the effect of a therapeutic change. 5) A consultation preparation module allows patients to indicate which topics they want to discuss during an outpatient visit. 6) Patients can ask for 'calling advise' if they are unsure whether to contact their physician. 7) Patients and healthcare providers can send each other text messages. 8) Interactive learning modules about PD. 9) Annual evaluation regarding patient satisfaction, self-management and healthcare consumption.

SUMMARY:
Introduction and rationale:

Parkinson´s disease (PD) is a slowly progressive and chronic disease, characterized by a range of motor and non-motor symptoms such as bradykinesia, tremor and falls, but also sleep disturbance, cognitive decline, behavioral problems and autonomic failure. These symptoms often fluctuate over time and between patients. These fluctuating and often debilitating symptoms necessitate proper monitoring. Due to this complexity, most patients require long-term specialized care. The current prevalence of PD in the Netherlands is estimated at 600-775 per 100.000 persons. This figure is expected to increase with > 50% in 2040. Combined with rising healthcare costs and a projected reduction in the number of available healthcare professionals, a system of frequent outpatient visits with a movement disorder specialist, as is currently the standard of care for PD in most (Dutch) hospitals, will likely not be sustainable.

Additionally, improvements can be made in the quality of care for PD-patients. The most important aspect mentioned by patients is improved self-management. Other points of improvement are: communication between different healthcare professionals involved; advanced care planning and having a single point of access / personal case manager. Recently an international group of experts in the field of PD have published a viewpoint article concerning their ideas for the optimization of the care for PD-patients. In addition to the previous points, these experts mention: providing care at home rather than in hospital; pro-active instead of reactive care and improvement of the expertise of healthcare professionals.

A possible solution to improving the sustainability of care for PD-patients, and addressing several of the issues concerning quality of care, lies in the use of telemedicine (or eHealth): the remote diagnosis and treatment of patients by means of telecommunications technology. Telemedicine exists in a wide variety of forms, one of which is 'telemonitoring'; the home monitoring of patients. In 2017 it was shown that telemonitoring is save and led to a significant reduction in health care consumption in patients with inflammatory bowel disease. Furthermore, studies in several chronic diseases have shown that telemonitoring leads to better patient empowerment and improved self-management. Self-management is in itself associated with improved health status and well-being in patients with a chronic disease as well as with a reduction in healthcare consumption.

In collaboration with Sananet, Zuyderland Medical Center has developed a telemonitoring tool for PD called 'SanaCoach Parkinson' (SCP). It is, to the investigators knowledge, the first telemonitoring tool for PD that uses anamnestic data from targeted questionnaires to monitor patients with PD. Trough the SCP both motor and non-motor aspects of PD are screened pro-actively. It allows patients to remain at home rather that visit the outpatient clinic. Additionally, proactive monitoring of symptoms leads to earlier detection of deterioration. This gives the neurologist the possibility to optimize (medical) treatment before further, costly, complications arise. Furthermore, the SCP improves patients' insight in their disease, supporting self-management.

A previous pilot-study into the effect of implementation of this tool showed that the use of the SCP was feasible in an outpatient care setting and that patient satisfaction and experienced quality of care were high. Additionally, the use of the SCP led to a significant reduction in the number of outpatient visits as well as the PD-related healthcare costs in Zuyderland Medical Center in the first year of use of the SCP.

Hypotheses:

The investigators hypothesize that implementation of telemonitoring via the SCP will be non-inferior to treatment as usual (TAU) with regards to the quality of care as experienced by PD-patients, while reducing the PD-related healthcare consumption and costs.

Secondly the investigators hypothesize that telemonitoring via the SCP will improve the quality of care for PD-patients compared to TAU.

Study Design and procedures:

This will be a non-randomized, prospective, multi-center, non-inferiority, implementation study. During 1 year, all consecutive PD-patients in the neurology outpatient clinic of each participating hospital that meet the in- and exclusion criteria will be invited to join this study. Participants will be monitored via the SCP for 2 years. During this time, PD-related outpatient visits with either a neurologist of specialized nurse will be set at 1-2 per patient per year, with a maximum total planned duration of 60 minutes. If this is not feasible, the primary reason for this will be recorded.

New hospitals may join the study until 6 months after the inclusion of the first patient.

Assessments will take place at baseline, 1 year and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis according to the Movement Disorder Society Clinical Diagnostic Criteria for Parkinson's Disease
* Disease duration ≥ 3 months.
* Able to complete the questionnaires and use the Sanacoach Parkinson, independently or with the help of an informal caregiver.

Exclusion Criteria:

* Not able to understand and/or sign the informed consent.
* No access to the internet via computer, tablet or smartphone.
* Participating in other trial

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-06-27 (Estimated)

PRIMARY OUTCOMES:
Patient-experienced quality of care | Change between baseline and after two years of using the Sanacoach Parkinson
  Measured by the net-promoter score. Each patient rates their care received on a scale of 0 to 10. Detractors (scoring 0-6) are subtracted from promoters (scoring 9-10), leaving the net-promoter score. The score ranges from -100 to +100, with higher scores indicating better patient-experienced quality of care.
Patient-satisfaction with the Sanacoach Parkinson | Measured after 2 years of using the Sanacoach Parkinson
  Measured by an 11-item patient satisfaction questionnaire. Score range = 1-45, with higher scores indicating better patient satisfaction.
Disease-related quality of life | Change between baseline and after two years of using the Sanacoach Parkinson
  Measured by the 8-item Parkinson's disease questionnaire (PDQ-8), range 0-32, higher scores indicate worse quality of life
Disease-related health care costs | Change of average costs per year during the two years of using the Sanacoach Parkinson, compared to a 6 month period before use of the Sanacoach Parkinson
  Calculated by measuring the number of PD-relates visits, telephone contacts and e-mail contacts with a neurologist, specialized nurse or general practitioner; number of hospitalizations, hospitalization days and emergency room visits related to PD, head trauma, hip fracture, pneumonia or psychosis; number of visits to a physiotherapist, occupational therapist, speech therapist or psychologist; number of days receiving inpatient of outpatient care at a rehabilitation center or nursing home; hours of formal and informal care received, days of labor missed and time spent by neurologists and specialized nurses on monitoring the Sanacoach Parkinson and follow-up activities. All these variables will be converted to costs per year (in euros).

SECONDARY OUTCOMES:
Patient self-management | Change between baseline and after two years of using the Sanacoach Parkinson
  Measured by the Partners In Health scale, range 0-96, higher scores indicate better self-management
Caregiver burden | Change between baseline and after two years of using the Sanacoach Parkinson
  Measured by the Caregiver Strain Index, range 0-13, higher scores indicate higher caregiver burden
Disease-severity | Change between baseline and after two years of using the Sanacoach Parkinson
  Measured by the Unified Parkinson's Disease Rating Scale (UPDRS), range 0-260, higher scores indicate increased disease-severity
Healthcare professional's attitude towards the Sanacoach Parkinson | Measured 6-monthly during 3 years of working with the Sanacoach Parkinson
  Measured by a 9-item questionnaire, range 0-36, higher scores indicate better satisfaction with the Sanacoach Parkinson

OTHER OUTCOMES:
Compliance with Sanacoach Parkinson | During the 2 years of using the Sanacoach Parkinson
  Number of periodic questionnaires completed, patients completing <3 questionnaires a year are defined as non-compliant
Number of patients requiring additional outpatient visits | During the 2 years of using the Sanacoach Parkinson
  % of patient years in which a patient requires more than 2 outpatient visits
Reasons for additional outpatient visits | During the 2 years of using the Sanacoach Parkinson
  Descriptive summary of the reasons patient required additional outpatient visits, as specified by healthcare providers. Pre-specified options are: 1) Doctor-initiated, physical examination needed 2) Doctor-initiated, deepen history 3) Doctor-initiated, nature of problem 4) Patient-initiated and 5) Caregiver-initiated

CONTACTS AND LOCATIONS:
Overall Officials: Gerrit Tissingh, MD, PhD, Principal Investigator — Zuyderland MC
Locations (6):
- Netherlands (6):
  - Meander Medical Center, Amersfoort
  - Onze Lieve Vrouwe Hospital, Amsterdam
  - Rode Kruis Hospital, Beverwijk
  - Zuyderland Medical Center, Geleen
  - Zuyderland Medical Center, Heerlen
  - Elkerliek Hospital, Helmond

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Poewe W, Seppi K, Tanner CM, Halliday GM, Brundin P, Volkmann J, Schrag AE, Lang AE. Parkinson disease. Nat Rev Dis Primers. 2017 Mar 23;3:17013. doi: 10.1038/nrdp.2017.13. PMID 28332488
- [Background] Clarke CE. Parkinson's disease. BMJ. 2007 Sep 1;335(7617):441-5. doi: 10.1136/bmj.39289.437454.AD. No abstract available. PMID 17762036
- [Background] Willis AW, Schootman M, Evanoff BA, Perlmutter JS, Racette BA. Neurologist care in Parkinson disease: a utilization, outcomes, and survival study. Neurology. 2011 Aug 30;77(9):851-7. doi: 10.1212/WNL.0b013e31822c9123. Epub 2011 Aug 10. PMID 21832214
- [Background] Willis AW, Schootman M, Tran R, Kung N, Evanoff BA, Perlmutter JS, Racette BA. Neurologist-associated reduction in PD-related hospitalizations and health care expenditures. Neurology. 2012 Oct 23;79(17):1774-80. doi: 10.1212/WNL.0b013e3182703f92. Epub 2012 Oct 10. PMID 23054239
- [Background] Kowal SL, Dall TM, Chakrabarti R, Storm MV, Jain A. The current and projected economic burden of Parkinson's disease in the United States. Mov Disord. 2013 Mar;28(3):311-8. doi: 10.1002/mds.25292. Epub 2013 Feb 21. PMID 23436720
- [Background] Vlaanderen FP, Rompen L, Munneke M, Stoffer M, Bloem BR, Faber MJ. The Voice of the Parkinson Customer. J Parkinsons Dis. 2019;9(1):197-201. doi: 10.3233/JPD-181431. PMID 30373962
- [Background] Bloem BR, Henderson EJ, Dorsey ER, Okun MS, Okubadejo N, Chan P, Andrejack J, Darweesh SKL, Munneke M. Integrated and patient-centred management of Parkinson's disease: a network model for reshaping chronic neurological care. Lancet Neurol. 2020 Jul;19(7):623-634. doi: 10.1016/S1474-4422(20)30064-8. Epub 2020 May 25. PMID 32464101
- [Background] de Jong MJ, van der Meulen-de Jong AE, Romberg-Camps MJ, Becx MC, Maljaars JP, Cilissen M, van Bodegraven AA, Mahmmod N, Markus T, Hameeteman WM, Dijkstra G, Masclee AA, Boonen A, Winkens B, van Tubergen A, Jonkers DM, Pierik MJ. Telemedicine for management of inflammatory bowel disease (myIBDcoach): a pragmatic, multicentre, randomised controlled trial. Lancet. 2017 Sep 2;390(10098):959-968. doi: 10.1016/S0140-6736(17)31327-2. Epub 2017 Jul 14. PMID 28716313
- [Background] Wilde MH, Garvin S. A concept analysis of self-monitoring. J Adv Nurs. 2007 Feb;57(3):339-50. doi: 10.1111/j.1365-2648.2006.04089.x. PMID 17233653
- [Background] Qian W, Lam TT, Lam HHW, Li CK, Cheung YT. Telehealth Interventions for Improving Self-Management in Patients With Hemophilia: Scoping Review of Clinical Studies. J Med Internet Res. 2019 Jul 10;21(7):e12340. doi: 10.2196/12340. PMID 31293241
- [Background] Jalil S, Myers T, Atkinson I. A meta-synthesis of behavioral outcomes from telemedicine clinical trials for type 2 diabetes and the Clinical User-Experience Evaluation (CUE). J Med Syst. 2015 Mar;39(3):28. doi: 10.1007/s10916-015-0191-9. Epub 2015 Feb 13. PMID 25677954
- [Background] Barlow J, Wright C, Sheasby J, Turner A, Hainsworth J. Self-management approaches for people with chronic conditions: a review. Patient Educ Couns. 2002 Oct-Nov;48(2):177-87. doi: 10.1016/s0738-3991(02)00032-0. PMID 12401421
- [Background] Lorig KR, Holman H. Self-management education: history, definition, outcomes, and mechanisms. Ann Behav Med. 2003 Aug;26(1):1-7. doi: 10.1207/S15324796ABM2601_01. PMID 12867348
- [Background] Allegrante JP, Wells MT, Peterson JC. Interventions to Support Behavioral Self-Management of Chronic Diseases. Annu Rev Public Health. 2019 Apr 1;40:127-146. doi: 10.1146/annurev-publhealth-040218-044008. Epub 2019 Jan 2. PMID 30601717
- [Background] Bodenheimer T, Lorig K, Holman H, Grumbach K. Patient self-management of chronic disease in primary care. JAMA. 2002 Nov 20;288(19):2469-75. doi: 10.1001/jama.288.19.2469. PMID 12435261
- [Background] Jie L, Jie A, Hoff J, Tissingh G. Telemonitoring verbetert parkinsonzorg. Medisch Contact. 2016; 14:7
- [Background] Wijers A, Hochstenbach L, Tissingh G. Telemonitoring via Questionnaires Reduces Outpatient Healthcare Consumption in Parkinson's Disease. Mov Disord Clin Pract. 2021 Jul 19;8(7):1075-1082. doi: 10.1002/mdc3.13280. eCollection 2021 Oct. PMID 34631943
- See also: Information on the epidemiology of Parkinson's Disease in the Netherlands, from the 'Rijksinstituut voor Volksgezondheid en Milieu' (RIVM), the Dutch National Institute for Health and Environment — https://www.volksgezondheidenzorg.info/onderwerp/ziekte-van-parkinson/cijfers-context/huidige-situatie
- See also: Report on demographic changes in the Netherlands from 2010 to 2040, by the 'Planbureau voor de Leefomgeving', the Dutch national institute for strategic policy analysis in the field of environment, nature and space — https://www.pbl.nl/sites/default/files/downloads/PBL_2013_Demografische_ontwikkelingen-2010-2040_1044.pdf